CLINICAL TRIAL: NCT03943524
Title: Evaluation of a Drug Interactions Software (Interax-AI) in Outpatients.
Brief Title: Drug Interactions in Outpatients.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties during the COVID pandemic
Sponsor: University of Buenos Aires (Other)
Collaborators: DrApp S.A. (Unknown)
Responsible Party: Principal Investigator, Guillermo Alberto Keller, Head of Pharmacovigilance Program, University of Buenos Aires
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RB-002
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Polypharmacy; Outpatient; Drug Interaction; Adverse Drug Reaction
Keywords: Polypharmacy; Outpatient; Drug Interaction; Adverse Drug Reaction; DrApp; Interax-AI
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Allocation: Non-Randomized An electronic medical record, DrApp, will be used, which will include a drug interaction program, Interax-AI, which will automatically indicate the medication prescriptions that involve a risk for the patient.
  All indications of each outpatient will be registered. The indications will be compared in the 4 months prior to the incorporation of the Interax-AI program with the 4 months after the incorporation of the program. Between both stages a period of 2 weeks will be established in which the data will not be recorded. The minimum number of patients that will be included in each stage is 100 and the maximum 200.
  Masking: Triple (Participant, Care Provider, Investigator) Primary Purpose: Prevention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DrApp Without Interax-AI (No Intervention): There are approximately 100 outpatients in whom the indications were registered through the use of DrApp, before the implementation of the drug interactions detection module.
- DrApp With Interax-AI (Experimental): There are approximately 100 outpatients in whom the indications were registered through the use of DrApp, AFTER the implementation of the drug interactions detection module (Interax-AI).
  Intervention: Device: Medication Interaction System of Dr App (Interax-AI)
  Interventions: Device: Interax-AI

INTERVENTIONS:
Device: Interax-AI — Interax-AI is a drug interactions detection module for the electronic clinical history software DrApp
  Arms: DrApp With Interax-AI

SUMMARY:
Multiple morbidity is increasing, especially in elderly people, with a corresponding increase in polypharmacy and inappropriate prescriptions. According to different evaluations, between 25 and 75% of patients aged 75 or older are exposed to 5 or more drugs. There is increasing evidence that polypharmacy can cause more harm than good, especially in elderly people, due to factors such as drug-drug and drug-disease interactions.

Many strategies were proposed to reduce polypharmacy and inappropriate prescribing, but there is little evidence to show benefit. There is an urgent need to implement effective strategies. The application methodology must be simple so that it does not fail in daily practice.

For the current plan, an electronic medical record, named "DrApp", will be used, which will include a drug interaction program, (Interax-AI), which will automatically indicate the medication prescriptions that involve a risk for the patient.

All outpatient indications followed by physicians using the DrApp electronic history will be registered. The indications will be compared in the 4 months prior to the incorporation of the Interax-AI program with the 4 months after the incorporation of the program. Between both stages a period of 2 weeks will be established in which the data will not be recorded. The minimum & maximum number of patients that will be included in each stage are 100 & 200.

The primary end point is to compare the total number of indications per inpatient, before the availability of the Interax-AI program and after the application of this program.

The objective is to evaluate if the computer program of detection of drug interactions allows to limit the polypharmacy in outpatients.

DETAILED DESCRIPTION:
Multiple morbidity is increasing, especially in elderly people, with a corresponding increase in polypharmacy and inappropriate prescriptions. According to different evaluations, between 25 and 75% of patients aged 75 or older are exposed to 5 or more drugs. There is increasing evidence that polypharmacy can cause more harm than good, especially in elderly people, due to factors such as drug-drug and drug-disease interactions.

Many strategies were proposed to reduce polypharmacy and inappropriate prescribing, but there is little evidence to show benefit. There is an urgent need to implement effective strategies. The application methodology must be simple so that it does not fail in daily practice.

For the current plan, an electronic medical record, named "DrApp", will be used, which will include a drug interaction program, (Interax-AI), which will automatically indicate the medication prescriptions that involve a risk for the patient.

All outpatient indications followed by physicians using the DrApp electronic history will be registered. The indications will be compared in the 4 months prior to the incorporation of the Interax-AI program with the 4 months after the incorporation of the program. Between both stages a period of 2 weeks will be established in which the data will not be recorded. The minimum & maximum number of patients that will be included in each stage are 100 & 200.

The primary end point is to compare the total number of indications per inpatient, before the availability of the Interax-AI program and after the application of this program.

The objective is to evaluate if the computer program of detection of drug interactions allows to limit the polypharmacy in outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients followed in outpatient clinics of doctors using the electronic medical record application DrApp

Exclusion Criteria:

* Lack of registration of medications used by the patient in the DrApp application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of polypharmacy cases detected in outpatients of outpatient clinics of doctors using the electronic medical record application DrApp | 1 year
  Through the electronic medical record called DrApp, the quantity of medicines prescribed to each patient is quantified and used for calculation of polypharmacy prevalence in tha basal period (pre-introduction of Interax-AI) and late period (Post introduction of Interax-AI).

SECONDARY OUTCOMES:
Interax-AI associated change in the number of total prescribed drug per patient | 1 year
  Change in total prescribed drug per patient will be calculated as the differene between basal total prescribed drug per patient (Pre-Interax-AI) minus resulting total prescribed drug per patient (Post-Interax-AI)
Number of total drug interactions per patient and subclassification by severity (in post-Interax-AI period). | 1 year
  The addition of the application called Interax-AI, will allow detecting the presence of drug interactions and their severity in the second phase. These will be reported as the total number of interactions reported per patient, and subclassificated into number of mild (no need to take action), moderate (require patient monitoring), and severe (possible contraindication) interactions detected per patient.
Difference between Number of total drug interactions per patient in the local environment with those reported in the literature at the international level. | 1 year
  The difference will be calculated as the number of total drug interactions per patient minus the value (number of drug interaction per patient) reported in the bibliography at international level in similar populations.

CONTACTS AND LOCATIONS:
Locations (3):
- Argentina (3):
  - Hospital de Clínicas José de San Martín, Buenos Aires, Buenos Aires F.D.
  - Centro de Vigilancia y Seguridad de Medicamentos, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.
  - Instituto de Investigaciones Cardiológicas Prof. Dr. Alberto C. Taquini, Ciudad Autonoma de Buenos Aire, Buenos Aires F.D.

IPD SHARING:
Plan to Share IPD: Yes
There is an intention to publish all the results obtained and share them with other researchers.
Supporting Information: Study Protocol, ICF
Time Frame: 1 Year